CLINICAL TRIAL: NCT05360121
Title: Effects of Muscle Energy Technique and General Stretching in the Management of Sub-acute Non-specific Low Back Pain :A Randomized Control Trial
Brief Title: Muscle Energy Technique Versus Back Stretching Among Non-specific Low Back Pain-subacute
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Abdul Rehman, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARehman
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Hyperthermia, Induced

STUDY DESIGN:
Intervention Model Description: Single blinding will be used in which only the researcher doing the study knows which treatment or intervention the participant is receiving until the trial is over.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique+ Thermotherapy +Back Strengthening exercise (Experimental)
  Interventions: Other: Muscle energy technique of erector spinae muscle; Other: Muscle energy technique of quadratus lumborum muscle; Other: Back strengthening exercises; Other: Thermotherapy
- General stretching+ Thermotherapy +Back Strengthening exercise (Active Comparator)
  Interventions: Other: Stretching of erector spinae muscle; Other: Stretching of quadratus lumborum muscle; Other: Back strengthening exercises; Other: Thermotherapy

INTERVENTIONS:
Other: Muscle energy technique of erector spinae muscle — Therapist will develop cross hand position left hand on lower thoracic and right hand on sacrum. Patient will asked to lift shoulder out of couch to contract the lumber erector spinae and apply force twenty percent against therapist force and keep this position of muscle contraction 7 to 10 seconds then 5 second relax .
  Then therapist will take new position of muscle restriction by slacking and will hold 30 second that position at the end of restriction then will finally end stretch with three repetition. Muscle energy technique of erector spinae muscle.
  Arms: Muscle energy technique+ Thermotherapy +Back Strengthening exercise
Other: Muscle energy technique of quadratus lumborum muscle — Therapist will take step over the patient off leg and squeezes gently with their thigh. Patient will abduct leg with 20 percent force against the resistance of therapists thigh for 7 to 10 second. the therapist gently and passively will move patient leg towards adduction by squatting down slowly. Therapist at same time with both hands cradling the iliac crest of pelvic for 30 second stretch and 3 repetition.
  Arms: Muscle energy technique+ Thermotherapy +Back Strengthening exercise
Other: Stretching of erector spinae muscle — The therapist standing on the side in a way to place his elbow placed on erector spine and apply stretching on the muscle belly in the direction of longitudinal or transverse plane( figure 1).Duration of stretch will be 15 seconds and four repetition.
  Arms: General stretching+ Thermotherapy +Back Strengthening exercise
Other: Stretching of quadratus lumborum muscle — Placing patient's legs to one side of the table and upper body also move to the same side in lateral flexion. This position generate a basic gentle stretch of the muscle. The therapist use elbow on tight/ flat part of muscle belly to stretch out the muscle(figure 2). Duration of stretch will be 15 seconds and four repetition
  Arms: General stretching+ Thermotherapy +Back Strengthening exercise
Other: Back strengthening exercises — 1. Supine Abdominal Draw In
  2. Supine Butt Lift with Arms at Side
  3. Abdominal Draw In with Heel Slide
  4. Abdominal Draw In with Knee to Chest
  5. Abdominal Draw In with feet on the ball
  6. Abdominal Draw In with feet on the ball- add movement
Other: Thermotherapy — Ten minute duration of hot pack given on low back for local superficial heat.

SUMMARY:
This study will highlight LBP management using MET and stretching application among subacute type of back pain

DETAILED DESCRIPTION:
This study will explore effects of two approaches , out of two MET has not been used in clinical practice more often, therefore this study will explore its physiological impact among back pain

ELIGIBILITY:
Inclusion Criteria:

- low back pain (subacute)

* VAS score( more than 3 cm)
* Quadratus lumborum and erector spinae tightness present

Exclusion Criteria:

* back pain (specific)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Visual Analogue scale scores at 3 weeks | at baseline and 3 weeks
  It is subjective outcome measure for pain intensity on 1 to10 cm scores. The '0 cm' score refers no pain and '10 cm' refers more excruciating pain. Increase in scores suggest worst pain intensity.
Change from Rolland Morris Disability Questionnaire scores at 3 weeks | at baseline and 3 weeks
  It is explore area of function leading to understand the level of disability. It consists of total 24 scores. The '0' score refers no disability and '24' refers maximum disability. Increase in scores suggest worst disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of physical medicine and rehabilitation, Karachi, Sindh, Pakistan